CLINICAL TRIAL: NCT03215147
Title: Prevalence and Impact on Quality of Life of Airway Disease in Patients With Idiopathic Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun Mi Choi, Assistant professor, Seoul National University Hospital
Other Study IDs: ILD Asthma
Record Dates: First submitted 2017-06-18; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Idiopathic Pulmonary Fibrosis; Airway Disease
Keywords: Idiopathic Pulmonary Fibrosis; Airway Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Confirmation of Airway Disease combined with IPF — To confirm the airway disease combined with IPF, PFT+BDR+DLCO, MBPT, Induced sputum exam, MAST, Total IgE, serum Eosinophil count, FENO will be done at the time of registration and 6~8 weeks later.

SUMMARY:
The investigators assess the prevalence of airway disease associated with idiopathic pulmonary fibrosis in Korea, and evaluate the effect of these airway diseases on the symptoms and quality of life of patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is defined as a specific form of chronic, progressive fibrosing interstitial pneumonia of unknown cause, occurring primarily in older adults, and limited to the lungs. It is characterized by progressive worsening of dyspnea and lung function and is associated with a poor prognosis.

The main symptoms of patients with IPF are dyspnea on exertion and a persistent dry cough or mildly productive cough.

In many IPF patients, cough is often the first symptom, preceding dyspnea on exertion sometimes by years. It affects upwards of 70-85% of patients with IPF.

Chronic obstructive pulmonary disease (prevalence rate 4-18%) and asthma (prevalence rate 5.9-9.9%) are the airway disease whose main symptoms are also dyspnea and cough.

To date, the effect of airway disease has not been well studied in patients with idiopathic pulmonary fibrosis, and the prevalence is unknown in Korea.

Unlike idiopathic pulmonary fibrosis, airway disease is a treatable, modifiable disease, so treatment of these diseases may improve QOL in IPF patients.

Therefore, this study's purpose is A. Identify the prevalence of airway disease in IPF patients B. Identify differences in QOL and symptoms according to presence of airway disease C. Identify the symptomatic improvement after active treatment for the airway diseases

ELIGIBILITY:
Inclusion Criteria:

* IPF patients

Exclusion Criteria:

* Patients on systemic steroid
* Patients with acute exacerbation within the last 6 months
* PFT+BDR, MBPT contra-indication
* SpO2 < 90%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ILD registry(Seoul National University IRB, IRB No. 1312-048-542), outpatient department, ward
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have asthma combined with idiopathic pulmonary fibrosis | Through study completion, an average of 2 year
  Confirmation of asthma : pulmonary function test with bronchodilator response or Methacholine provocation test
Number of participants who have COPD combined with idiopathic pulmonary fibrosis | Through study completion, an average of 2 year
  Confirmation of COPD : pulmonary function test with bronchodilator response
Number of participants who have Eosinophilic bronchitis combined with idiopathic pulmonary fibrosis | Through study completion, an average of 2 year
  Confirmation of Eosinophilic bronchitis : pulmonary function test with bronchodilator response, induced sputum

SECONDARY OUTCOMES:
The difference of CAT scores between patients with airway disease and those without airway disease. | baseline and after treating the airway disease for 6~8 weeks
  Quality of life : COPD assessment test(CAT)
The difference of SGRQ scores to assess quality of life between patients with airway disease and those without airway disease. | baseline and after treating the airway disease for 6~8 weeks
  Quality of life : St George's Respiratory Questionnaire(SGRQ)
The difference of mMRC scores to assess symptom severity between patients with airway disease and those without airway disease. | baseline and after treating the airway disease for 6~8 weeks
  Symptom severity : mMRC
The difference of distance of 6MWT to assess symptom severity between patients with airway disease and those without airway disease. | baseline and after treating the airway disease for 6~8 weeks
  Symptom severity : 6 minute walking test(6MWT)
The difference of EQ-5D-VAS scores to assess symptom severity between patients with airway disease and those without airway disease. | baseline and after treating the airway disease for 6~8 weeks
  Symptom severity : EQ-5D-VAS
The difference of CQLQ scores to assess symptom severity between patients with airway disease and those without airway disease. | baseline and after treating the airway disease for 6~8 weeks
  Symptom severity : Cough Quality-of-Life Questionnaire(CQLQ)
Checking the improvement of CAT score to assess the quality of life between patients with airway disease and those without airway disease | After treating the airway disease for 6~8 weeks
  Quality of life : COPD assessment test(CAT)
Checking the improvement of SGRQ score to assess the quality of life between patients with airway disease and those without airway disease | After treating the airway disease for 6~8 weeks
  Quality of life : St George's Respiratory Questionnaire(SGRQ)
Checking the improvement of mMRC scores to assess symptom severity between patients with airway disease and those without airway disease | After treating the airway disease for 6~8 weeks
  Symptom severity : mMRC
Checking the improvement of distance of 6MWT to assess symptom severity between patients with airway disease and those without airway disease | After treating the airway disease for 6~8 weeks
  Symptom severity : 6 minute walking test(6MWT)
Checking the improvement of EQ-5D-VAS score to assess symptom severity between patients with airway disease and those without airway disease | After treating the airway disease for 6~8 weeks
  Symptom severity : EQ-5D-VAS
Checking the improvement of CQLQ to assess symptom severity between patients with airway disease and those without airway disease | After treating the airway disease for 6~8 weeks
  Symptom severity : Cough Quality-of-Life Questionnaire(CQLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Choi Sun Mi, Principal Investigator — Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine and Lung institute, Seoul National University College of Medicine, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea